CLINICAL TRIAL: NCT04835428
Title: A Randomized, Single-Blinded, Non-Inferiority Study Comparing AGN1 Local Osteo-Enhancement Procedure (LOEP) SV Kit Treatment of Vertebral Compression Fragility Fractures to PMMA Bone Cement Treatment
Brief Title: STAND - Study of the AGN1 LOEP SV Kit Compared to PMMA in Patients With Vertebral Compression Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AgNovos Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGN-CIP-201; STAND (Other: AgNovos)
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Vertebral Compression Fracture; Compression Fracture; Vertebral Compression
Keywords: LOEP; AGN1; STAND; Local Osteo-Enhancement Procedure
MeSH Terms: conditions — Fractures, Compression

STUDY DESIGN:
Intervention Model Description: Four hundred eight (408) eligible subjects at up to twenty-five (25) study sites will be randomized 1:1 for treatment using the AGN1 LOEP SV Kit (Intervention Group) or PMMA bone cement (Active Control Group).
Who Masked: Participant
Masking Description: Study subjects will not be informed of their treatment group assignment at the time of randomization or at any time before the subject's last office visit. The blind will be broken only if it is necessary to protect the safety or welfare of the subject as determined by the Investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment with AGN1 LOEP SV Kit (Experimental): The AGN1 LOEP SV Kit is intended for fixation of pathological fractures of the vertebral body using vertebral augmentation. Following saline lavage to create space, the AGN1 implant material is injected and hardens in situ to augment the fractured vertebral body. The AGN1 implant material is then resorbed and replaced with new bone.
  Interventions: Device: Treatment Group: AGN1 LOEP SV Kit
- Treatment with PMMA bone cement (Active Comparator): High viscosity PMMA bone cement will be used for vertebral augmentation.
  Interventions: Device: Control Group: PMMA bone cement

INTERVENTIONS:
Device: Treatment Group: AGN1 LOEP SV Kit — The AGN1 LOEP SV Kit is intended for fixation of pathological fractures of the vertebral body using vertebral augmentation. Following saline lavage to create space, the AGN1 implant material is injected and hardens in situ to augment the fractured vertebral body. The AGN1 implant material is then resorbed and replaced with new bone.
  Arms: Treatment with AGN1 LOEP SV Kit
Device: Control Group: PMMA bone cement — High viscosity PMMA bone cement will be used for vertebral augmentation.
  Arms: Treatment with PMMA bone cement

SUMMARY:
This is a multicenter, single-blinded, randomized controlled clinical trial evaluating the safety and efficacy of the AGN1 LOEP SV Kit for the treatment of painful vertebral compression fragility fractures (VCFs). The objective of this study is to demonstrate non-inferiority of the AGN1 LOEP SV Kit for the treatment of VCFs to standard of care vertebroplasty treatment using bipedicular injection of PMMA bone cement.

DETAILED DESCRIPTION:
Four hundred and eight (408) eligible subjects at up to twenty-five (25) study sites will be randomized 1:1 for treatment using the AGN1 LOEP SV Kit (Intervention Group) or PMMA bone cement (Active Control Group).

1. Intervention Group - receives vertebral augmentation of the target VCF(s) using the AGN1 LOEP SV Kit
2. Active Control Group - receives vertebral augmentation of the target VCF(s) using either Stryker VertaPlex HV or Medtronic Kyphon HV-R.

Follow-up visits will be conducted at 7 days, 28 days, 3 months, 12 months and 24 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female 50 years of age or older at the time of study treatment.
2. Subject has one (1) or two (2) acute VCF(s). Note that subjects are eligible if they have an asymptomatic, healed VCF(s) at any non-target vertebral level.
3. Each target VCF meets all of the following criteria:

   1. Due to diagnosed or presumed underlying osteoporosis
   2. T1 to L5 inclusively
   3. Target VCF-related pain ≤ 6 months at time of study treatment
4. Each target VCF shows loss of height of the vertebral body ≤ 50% based on X-ray at baseline.
5. Each target VCF is acute or persistent (not healed), as demonstrated on imaging, including T2-weighted, STIR MRI, bone scan or bone scan with SPECT/CT, serial radiographs, or other serial imaging demonstrating acuity.
6. Focal tenderness to palpation of the spinal process of each target VCF on the physical exam correlates with imaging.
7. Subject has failed conservative medical therapy (bed rest, observation, chiropractic care, orthotics, opioid and non-opioid analgesics, and/or physical therapy), defined as either having a VAS back pain score of ≥ 70 mm after 24 hours to 6 weeks of conservative care or a VAS back pain score of ≥ 50 mm after more than 6 weeks of conservative care.
8. Subject has an Oswestry Disability Index (ODI) score of ≥ 30% at baseline.
9. Subject is capable of giving written informed consent to participate in the study.
10. The subject's willingness, ability, and commitment to participate in screening, treatment, and all follow-up evaluations for the full length of the study has been documented

Exclusion Criteria:

1. At least one of the target VCF(s) is unstable, including split or burst fracture.
2. Subject has a bleeding disorder.
3. Subject has an active infection of the spine or surgical site.
4. Subject has a bloodborne infection.
5. At least one of the target VCFs is due to underlying or suspected tumor.
6. At least one of the target VCFs is due to high-energy trauma.
7. At least one of the target VCFs is due to osteonecrosis.
8. At least one of the target VCFs has a local kyphotic angle of > 30 degrees, measured as the angle between the superior endplate and inferior endplate at the target VCF.
9. Subject has had any prior surgical treatment at the target vertebral level or adjacent vertebral levels.
10. The pedicle(s) in the target vertebral body appears unable to safely accommodate transpedicular access instrumentation.
11. Subject has neurologic symptoms, deficits, or radiculopathy related to the target VCF(s).
12. Subject has spinal canal compromise causing clinical manifestations of cord, neural foramen, or nerve root compression at the level to be treated.
13. Subject has pain, progressive weakness, or paralysis due to herniated nucleus pulposus or spinal stenosis.
14. Subject has spondylolisthesis > Grade 1 at target vertebral body(ies).
15. Subject requires daily opioid medication for pain not related to the target VCF(s).
16. Subject has severe cardiopulmonary deficiencies.
17. Subject has a Body Mass Index (BMI) > 35.
18. Subject has a history of metabolic bone disease other than osteoporosis (e.g., Paget's disease, renal osteodystrophy, or osteomalacia).
19. Subject has a history of tuberculous spondylitis.
20. Subject has a history of invasive malignancy within the last five (5) years, other than non-melanoma skin cancer. Subject is not excluded if they have a history of malignancy over 5 years ago treated with curative intent and without clinical signs or symptoms since then.
21. Subject is on oral or parenteral immune-suppressive drugs.
22. Subject has uncontrolled diabetes mellitus.
23. Subject has severe renal insufficiency defined as an estimated glomerular filtration rate (eGFR) < 30 mL/min.
24. Subject has a diagnosed calcium metabolism disorder.
25. Subject has known allergies to calcium-based bone void fillers.
26. Subject is pregnant or planning to become pregnant during participation in the study.
27. In the judgment of the Investigator, the subject is not a good study candidate. (e.g. substance abuse or chemical dependency, inability to adhere to follow-up schedule, progression of the fracture between screening and the procedure visit).
28. Subject is currently enrolled in another interventional clinical study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in VCF-related Pain as measured by a 100 mm Visual Analogue Scale (VAS) | 24 months
  Change in VCF-related pain by > 20 mm from baseline as measured by a 100 mm Visual Analogue Scale (VAS) where 0mm is no pain, and 100mm is worst pain possible.
Change in function | 24 months
  change of function from baseline as measured by the Oswestry Disability Index (ODI)
Radiographic evidence of implant resorption (Intervention Group only) | 24 months
  change in resorption from procedure as assessed by independent radiographer
Radiographic evidence of bone formation (Intervention Group only) | 24 months
  change in bone formation from procedure as assessed by independent radiographer
Adverse events | 24 months
  Occurrence of device-related serious adverse events, device-related adverse events or serious adverse events categorized as failure or surgical intervention at the target level occurring post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kern Singh, Principal Investigator — Midwest Orthopedics at Rush
Locations (19):
- United States (19):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Elite Pain and Spine Institute, Mesa, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Orlando Neurosurgery (Conquest Research), Orlando, Florida
  - Cleveland Clinic Florida, Stuart, Florida
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Duly Health / NextStage Clinical Research, Naperville, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Abay Neuroscience Center / NextStage Clinical Research, Wichita, Kansas
  - Louisiana Spine Institute, Shreveport, Louisiana
  - Anne Arundel Medical Center (AAMC), Annapolis, Maryland
  - Lahey Medical Center, Burlington, Massachusetts
  - Washington University St. Louis, St Louis, Missouri
  - Mt. Sinai, New York, New York
  - Montefiore, The Bronx, New York
  - Pinehurst Surgical Clinic, Pinehurst, North Carolina
  - Texas Back Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No